CLINICAL TRIAL: NCT02031445
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of MRX-6 Cream 2% in Pediatric Subjects With Mild to Moderate Atopic Dermatitis Followed by an Open Label Extension
Brief Title: Double-Blind, Trial to Evaluate the Safety and Efficacy of MRX-6 Cream 2%
Acronym: C012013
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis showed lack of efficacy
Sponsor: Celsus Therapeutics PLC (Industry)
Responsible Party: Sponsor
Organization: AKARI Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C012013
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): BID
  Interventions: Other: Placebo
- MRX-6 (Experimental): BID
  Interventions: Drug: MRX-6

INTERVENTIONS:
Drug: MRX-6
  Arms: MRX-6
Other: Placebo
  Arms: Placebo

SUMMARY:
Randomized, double-blind, parallel group, placebo-controlled, multicenter, efficacy and safety study in subjects with mild to moderate atopic dermatitis.

Following the double blind period, subjects will be allowed to continue treatment with topical MRX-6 Cream 2% in an open-label extension. Demonstrate the efficacy of MRX-6 Cream 2% compared to Vehicle for the treatment of the signs and symptoms of atopic dermatitis and demonstrate the safety of MRX-6 Cream 2% for the treatment of the signs and symptoms of atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, ≥2 years of age and ≤17 years of age, of any race or ethnicity
* Must have clinical diagnosis of mild to moderate atopic dermatitis (AD) at both Screening and Baseline Visits, defined as IGA score of 2 or 3 (Hanifin and Rajka, Rothe 1980)
* Must have AD affecting ≥ 5% total body surface area (TBSA) at Baseline
* History of AD for at least 3 months prior to Baseline
* Informed consent/assent in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guideline (21 CFR §50.25[c]) and applicable regulations, before completing any study-related procedures

Exclusion Criteria:

* Use of topical corticosteroids within 7 days prior to Baseline
* Use of systemic corticosteroids, topical calcineurin inhibitors, photo-therapy (eg, PUVA, UVB) or immunosuppressive therapy (eg, cyclosporine) within 14 days prior to Baseline
* Subjects that require systemic therapy for the treatment of atopic dermatitis
* Use of systemic anti-infective or antibiotic treatment within 14 days prior to Baseline
* Subjects who present with clinical conditions other than AD that may interfere with the evaluation (eg, generalized erythroderma, acne, Netherton's Syndrome, psoriasis)
* Secondary infection of AD (bacterial, viral or fungal) within the skin area under study or open skin infections in any area at Baseline
* Women of childbearing potential who are lactating or pregnant as determined by urine pregnancy test at Screening. • History of MRX-6 cream 2% sensitivity or to any component of the test article
* History of severe anxiety and/or depression; any history of suicide attempt
* Subjects with a history of human immunodeficiency virus (HIV) as determined by medical history
* Subjects with any screening clinical laboratory result outside the normal range that is clinically relevant in the opinion of an appropriately qualified physician
* Subjects who, in the opinion of the Investigator, would be non compliant with the visit schedule or study procedures
* Participation in any other investigational trial within 6 weeks of Baseline, or during study conduct
* Chronic condition(s) which are either unstable or not adequately controlled
* Use of non-sedating anti-histamines within 7 days of first dose or at any time during study conduct
* Drug or alcohol abuse, mental dysfunction, or other condition limiting the subject's ability to be compliant with study-related procedures

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment | 4 weeks

SECONDARY OUTCOMES:
Safety | 4 weeks
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Avner Shemer, Prof, Principal Investigator — Laniado Medical Center; Alex Zvulunov, Prof, Principal Investigator — Mayanei Hayeshua Medical Center; Eli Sprecher, Prof, Principal Investigator — Tel-Aviv Sourasky Medical Center; Dalia Gilat, Dr., Principal Investigator — Maccabi Healthcare Services, Israel; Lili Segal, Dr., Principal Investigator — Mayanei Hayeshua Medical Center; Jacob Mashiah, Dr., Principal Investigator — Dermatology Clinic, Tel Aviv, Kefar Saba
Locations (5):
- Israel (5):
  - Dermatology Clinic, Kfar Saba
  - Dermatology Clinic, Kiryat Ono
  - Lev Yasmin Clinic, Netanya
  - Dermatology Clinic, Petah Tikva
  - Sourasky Medical Center, Tel Aviv